CLINICAL TRIAL: NCT05226000
Title: Pharmacokinetics of Benaglutide Injection in Overweight/Obese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RH-RCT-IS-002
Record Dates: First submitted 2022-01-28; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Overweight/Obese Adults
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benaglutide Injection (Experimental): All subjects received multiple doses (tid) of 0.06 mg, 0.1 mg, 0.14 mg, and 0.2 mg in sequence, followed by the next dose after completing the previous multiple dosing. The administration time of each dose was 0.06 mg for 3 days, 0.1 mg for 3 days, 0.14 mg for 5 days, and 0.2 mg for 5 days.
  Interventions: Drug: Benaglutide Injection

INTERVENTIONS:
Drug: Benaglutide Injection — All subjects received multiple doses (tid) of 0.06 mg, 0.1 mg, 0.14 mg, and 0.2 mg in sequence, followed by the next dose after completing the previous multiple dosing. The administration time of each dose was 0.06 mg for 3 days, 0.1 mg for 3 days, 0.14 mg for 5 days, and 0.2 mg for 5 days.

SUMMARY:
This study is a open and multiple dose escalation phase I clinical study, aiming to evaluate the pharmacokinetic characteristics and safety of Benaglutide Injection in overweight/obese adults after multiple subcutaneous injections.

This study will enroll 16 overweight/obese adults, both male and female. The trial was divided into two batches, including 4 subjects who completed all dosing, safety assessment and telephone follow-up, and the remaining 12 subjects who were enrolled for the trial. All subjects received multiple doses (tid) of 0.06 mg, 0.1 mg, 0.14 mg, and 0.2 mg in sequence, followed by the next dose after completing the previous multiple dosing. The administration time of each dose was 0.06 mg for 3 days, 0.1 mg for 3 days, 0.14 mg for 5 days, and 0.2 mg for 5 days.

Subjects will be screened at D-14-D-2, and eligible subjects D-2 will be admitted to the phase I clinical trial ward at D-2. D-1 Blank blood samples were collected at different time points before and after breakfast for PK test baseline correction. D1 began by subcutaneously injecting different doses of benaglutide injection 5 minutes before the daily three meals, collecting biological samples at different time points after the first administration of D6, D7, D11, D12 and D16 to evaluate the pharmacokinetic characteristics of Benaglutide. Subjects will be discharged after all samples are collected and safety assessed at D17. Telephone follow-up was performed on the 7th day after discharge (D24±2) to further observe safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 70 years old (including the critical value).
* BMI meets the following requirements (a or b):

  1. BMI>28 kg/m2;
  2. BMI>24 kg/m2 with at least one of the following symptoms:

Vigorous appetite, hunger before meals unbearable, each meal into more food. Combined with hyperglycemia, hypertension, dyslipidemia, fatty liver in one or several.

Combined with weight-bearing joint pain. Obesity causes dyspnea or obstructive sleep apnea syndrome.

* The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: Vital signs, physical examination, blood routine, blood biochemistry, urinalysis, pregnancy test for female, serological tests for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), and syphilis virus, 12 lead ECG.
* The subjects have no family planning within 3 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* Patients with type 1 diabetes or type 2 diabetes with a clear diagnosis;
* Fasting intravenous blood glucose ≥7 mmol/L or 75g during screening. Oral glucose tolerance test (OGTT) two hours after glucose load;
* Fasting venous blood glucose <2.8 mmol/L at screening, and/or those with a history of hypoglycemia;
* Those who complained of a weight change of >5% within 3 months before screening;
* Have used weight loss drugs or hypoglycemic drugs that may affect body weight within 4 weeks before screening;
* Drugs used within 4 weeks before screening that may cause significant weight gain: including systemic glucocorticoid therapy (lasting more than 1 week); tricyclic antidepressants; antipsychotic or antidepressant drugs; may interfere with blood sugar regulation Functional medicine; all proprietary Chinese medicines and Chinese herbal medicines;
* Those who have a clear history of malignant tumors,
* People with Cushing's syndrome, hypothyroidism, polycystic ovary disease or other genetic endocrine diseases or medical history;
* Those who have a history of bariatric surgery;
* Have a history of multiple endocrine tumors or a family history; have a history of medullary thyroid carcinoma or other tumors, a family history;
* History of acute and chronic pancreatitis;
* Moderate to severe gastrointestinal diseases with additional gastrointestinal motility disorders or obstructive enteropathy;
* Have a clear history of mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 80 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 80 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 80 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞
elimination half-life time(T1/2) | 80 days
  Evaluation of elimination half-life time(T1/2)
The total clearance(CL) | 80 days
  Evaluation of the total clearance(CL)

SECONDARY OUTCOMES:
Incidence of Treatment Adverse Events | 80 days
  Collection of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China